CLINICAL TRIAL: NCT00769392
Title: Pilot Study: A Randomized Trial Of Anesthetic Agents For Intravitreal Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2008-076
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2019-03

CONDITIONS: Macular Degeneration
Keywords: Macular Degeneration; Intravitreal injections; Eye anesthesia-Topical/subconjunctival; Eye-surgical procedures; Ophthalmologic anesthesia methods
MeSH Terms: conditions — Macular Degeneration | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive a unique sequence of one of the 4 anesthetic agents per month, prior to a standard of care monthly intravitreal injection (1 injection per month for a total of 4 months). At the end of study participation, each patient will have received each of the 4 anesthetic agents once prior to one of the 4 intravitreal injections (ex. Randomization to sequence: Proparcacaine used prior to Injection 1; Tetracaine used prior to Injection 2; Lidocaine sponge used prior to Injection 3; Lidocaine suconjunctival injection used prior to Injection 4).
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Other): All Participants will be randomized to receive a unique sequence of one of the 4 anesthetic agents per month, prior to a standard of care monthly intravitreal injection (1 injection per month for a total of 4 months). At the end of study participation, each patient will have received each of the 4 anesthetic agents once prior to one of the 4 intravitreal injections (ex. Randomization to sequence: Proparacaine Ophthalmic drops used prior to Injection 1; Tetracaine Ophthalmic drops used prior to Injection 2; Lidocaine 4% sponge used prior to Injection 3; Lidocaine 2% injectable solution (subconjunctival) used prior to Injection 4).
  Interventions: Drug: Proparacaine Ophthalmic; Drug: Tetracaine Ophthalmic; Drug: Lidocaine 4%; Drug: Lidocaine 2% Injectable Solution

INTERVENTIONS:
Drug: Proparacaine Ophthalmic — Drops of Proparacaine on the eye, administered as described in the package insert
Drug: Tetracaine Ophthalmic — Drops of Tetracaine on the eye, administered as described in the package insert
Drug: Lidocaine 4% — A cotton sponge(pledget)soaked with Lidocaine 4% placed over the conjunctiva
Drug: Lidocaine 2% Injectable Solution — A subconjunctival injection of Lidocaine 2%

SUMMARY:
This study is designed to compare four currently used types of anesthesia used prior to intravitreal injection in order to evaluate the most effective method of anesthesia in reducing pain and discomfort associated with intravitreal injections.

DETAILED DESCRIPTION:
Over the last several years intravitreal injection of pharmacologic agents has become a common procedure in ophthalmology. Injected agents include steroid, antibiotics, and most recently anti-VEGF agents. There are many methods of preparing a patient for intravitreal injection. While there are guidelines for infection prophylaxis, there is currently no standard of care or consensus on which method of anesthesia is most effective in reducing pain and discomfort associated with intravitreal injections.

Patients who have received prior injections and are scheduled to continue regular injections will be randomized to utilize one of four types of anesthetic treatment for each of 4 treatment periods,so that each subject receives all four types of anesthesia over the course of the study. The order of the anesthetic treatment the subject will receive prior to each planned intravitreal injection during the study period will be different for each subject. This will decrease the effect of extraneous variables from influencing subjective pain scores.

Following each procedure, patients will fill out an analog pain scale questionnaire, grading the discomfort of receiving both the anesthesia and the injection(on separate 0-10 scales).

The anesthetic methods used will include: 1.) Drops of Proparacaine on the eye, 2.) Drops of Tetracaine on the eye, 3.) A cotton sponge (pledget) soaked with Lidocaine 4% placed over the conjunctiva and 4.)A subconjunctival injection with 2% Lidocaine.

The subjects' number and type of visits, tests and treatments will be standard of care and will not be different due to the study. The total time for the treatment part of the study coincides with four injections (1 injection per month) or approximately 4 months and will be followed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 40 years of age
* Diagnosis of age-related macular degeneration
* History of at least 1 intravitreal injection in the past in either eye
* Written informed consent has been obtained

Exclusion Criteria:

* Known allergy or sensitivity to the study medications(s), it's components, or other agents required for the study procedures(e.g. Povidone iodine)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08-12 (Actual); Study Completion 2009-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory R. Blaha, M.D., Ph.D., Principal Investigator — Lahey Clinic, Inc.
Locations (3):
- United States (3):
  - Lahey Clinic Arlington, Arlington, Massachusetts
  - Lahey Clinic, Inc., Burlington, Massachusetts
  - Lahey Clinic Northshore, Peabody, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaderli B, Avci R. Comparison of topical and subconjunctival anesthesia in intravitreal injection administrations. Eur J Ophthalmol. 2006 Sep-Oct;16(5):718-21. doi: 10.1177/112067210601600509. PMID 17061223
- [Background] Landry DA. Topical anesthetic pledgett system (TAPS) for intravitreal injection preparation. Insight. 2007 Oct-Dec;32(4):20. PMID 18306942

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 participants enrolled in this study. Once 24 subjects completed the study, the remaining 4 subjects were not required to complete the study, therefore, their data was not collected for this analysis.
Groups:
- All Study Participants: All participants received, in an randomized cross-over fashion, Proparacaine drops, Tetracaine drops, Lidocaine 4% soaked cotton sponge, and Lidocaine 2% subconjunctival injection.
Period: Overall Study
Arm/Group | All Study Participants
Started | 28
Completed | 24
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: 28 participants enrolled in this study. Once 24 subjects completed the study, the remaining 4 subjects were not required to complete the study and their data was not used in this analysis.
Groups:
- All Participants: Participants will be randomized to receive a unique sequence of one of the 4 anesthetic agents per month, prior to a standard of care monthly intravitreal injection (1 injection per month for a total of 4 months). At the end of study participation, each patient will have received each of the 4 anesthetic agents once prior to one of the 4 intravitreal injections (ex. Randomization to sequence: Proparcacaine used prior to Injection 1; Tetracaine used prior to Injection 2; Lidocaine sponge used prior to Injection 3; Lidocaine suconjunctival injection used prior to Injection 4).
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Discomfort Associated With the Intravitreal Injection
Description: Discomfort Associated With the Intravitreal Injection using a Subjective Analog Pain Scale (0-10); no pain (0) and severe pain (10)
Time Frame: 16 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 24
units on a scale
  Lidocaine 4% | 3 [0 to 9]
  Lidocaine 2% Injectable Solution | 2.3 [0 to 6]
  Proparacaine Ophthalmic | 2.8 [0 to 8]
  Tetracaine Ophthalmic | 3.1 [0 to 10]
Statistical Analysis 1: Comparison: All Participants; A comparison of injection discomfort using mean pain scores for all 4 anesthesia intervention agents used in this study; Test type: Other; p = 0.28, single factor analysis of variance

2. Secondary Outcome: Discomfort From Anesthesia Used Prior to Intravitreal Injections
Description: Discomfort from Anesthesia used prior to Intravitreal Injections using a Subjective Analog Pain Scale (0-10); no pain (0) and severe pain (10).
Time Frame: 16 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 24
units on a scale
  Lidocaine 4% | 1.4 [0 to 8]
  Lidocaine 2% Injectable Solution | 1.6 [0 to 6]
  Proparacaine Ophthalmic | 0.7 [0 to 8]
  Tetracaine Ophthalmic | 1.0 [0 to 4]
Statistical Analysis 1: Comparison: All Participants; A comparison of discomfort of all 4 anesthesia intervention agents used in this study using mean pain scores; Test type: Other; p = 0.17, single factor analysis of variance

ADVERSE EVENTS:
Time Frame: Adverse Event frequency was monitored from the time of participant consent to the end of the study at 6 months.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 13/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=24)
Subconjunctival Hemorrage with Lidocaine subconjunctival injection (Eye disorders) | 13 (13) — Subconjunctival Hemorrage occurrence with Lidocaine subconjunctival injection

LIMITATIONS AND CAVEATS:
Limitations of any study examining pain are the subjective nature of pain, the difficulty in measurement, and patient variability. This was address by using a randomized block design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes